CLINICAL TRIAL: NCT07059078
Title: PCORI Comparative Effectiveness Study: Comparative Effectiveness of Brief Motivational Interviewing +/- Adjunctive Smartphone App-delivered Mindfulness Training for Reducing Alcohol Use in Adolescents in Pediatric Primary Care Settings
Brief Title: Brief Motivational Interviewing +/- Mindfulness Training for Adolescent Alcohol Use in Pediatric Primary Care
Acronym: PCORIMINDSET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00452272
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Alcohol Use
Keywords: Alcohol use; Alcohol-related problems; Drug use; Adolescent; Motivational interviewing; Mindfulness; Mindfulness training; brief alcohol intervention; digital therapeutic intervention; SBIRT; PCORI
MeSH Terms: conditions — Underage Drinking; Alcohol Drinking | interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Care Provider
Masking Description: Research Assistant who is collecting patient data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Motivational interviewing-based Alcohol Intervention (BMAI) (Active Comparator): Participants randomized to this arm will receive a brief motivational interviewing-based alcohol intervention (BMAI) delivered in person by a pediatric clinician in the pediatric primary care (PPC) office setting.
  BMAI is adapted from the Provider Guide: Adolescent SBIRT Using the S2BI-CRAFFT Screening Tool and incorporates motivational interviewing (MI) principles. It includes clinician-delivered feedback, advice, and goal setting to help adolescents recognize links between alcohol/drug use and negative health outcomes, and to develop personalized change plans.
  BMAI is delivered across one or more visits, with the initial session typically lasting 10-30 minutes and follow-ups lasting 5-15 minutes. Clinicians delivering BMAI include pediatricians, nurses, and social workers who provide primary care to 12-17-year-olds at participating JHMI sites and who have completed SBIRT/BMAI training and monitoring as part of the trial.
  Interventions: Behavioral: Brief Motivational Interviewing-based Alcohol Intervention
- BMAI + Smartphone app-delivered Mindfulness Training (BMAI + MT) (Active Comparator): Participants randomized to this arm will receive the BMAI intervention described above plus 8 weeks of adjunctive smartphone-delivered mindfulness training (MT) via the Healthy Minds Program (HMP) app.
  The HMP app offers self-guided, self-paced mindfulness and meditation training, with core modules on Awareness, Insight, Connection, and Purpose. This study focuses on the Awareness and Insight modules, which teach breath and body awareness, noting of emotions, and the application of mindfulness in daily life.
  After randomization, participants will meet with study staff to download the app, receive instruction, and be asked to use it 5-30 minutes daily, following a pathway of 4 weeks of Awareness content, then 4 weeks of Insight content.
  After the 8-week MT period, participants will have open access to all HMP modules and be encouraged to explore the remaining content as desired during the follow-up period.
  Interventions: Behavioral: Brief Motivational Interviewing-based Alcohol Intervention; Behavioral: Smartphone App-delivered Mindfulness Training

INTERVENTIONS:
Behavioral: Brief Motivational Interviewing-based Alcohol Intervention — Participants in both arms (BMAI and BMAI + MT) will receive a brief motivational interviewing-based alcohol intervention (BMAI) delivered by a pediatric clinician in the primary care setting.
  BMAI is adapted from the Provider Guide: Adolescent SBIRT Using the S2BI-CRAFFT Screening Tool, grounded in the stages of change model and motivational interviewing (MI). It consists of one or more brief sessions involving structured feedback, advice, and goal setting to help adolescents recognize links between substance use and health outcomes and develop personalized change plans. The intervention is face-to-face, delivered during routine or follow-up visits, and modeled after the brief negotiated interview. The first session lasts 10-30 minutes and includes six MI-based steps. This is followed by one or more additional brief MI sessions lasting 5-15 minutes where the patient's goals are reviewed, gains or barriers are addressed, and ongoing support is provided.
Behavioral: Smartphone App-delivered Mindfulness Training — In addition to BMAI, participants in the BMAI + MT arm will receive 8 weeks of smartphone-delivered mindfulness training using the Healthy Minds Program (HMP) app.
  The HMP app provides self-guided, self-paced mindfulness and meditation training designed to improve psychological well-being, reduce stress/anxiety, and enhance self-regulation. It includes podcast-style teachings and guided meditations. The app features four modules-Awareness, Insight, Connection, and Purpose-based on neuroscience research. Each module offers 27 practices (5-30 minutes each). This study focuses on the Awareness and Insight modules, which teach breath and body awareness and emotion noting to support mindfulness in daily life. Participants will be asked to use the app 5-30 minutes per day, following 4 weeks of Awareness content, then 4 weeks of Insight. After 8 weeks, they will have open access to all modules and be encouraged to explore additional practices as they find helpful during follow-up.
  Arms: BMAI + Smartphone app-delivered Mindfulness Training (BMAI + MT)

SUMMARY:
Alcohol use is prevalent in U.S. adolescents and contributes to adverse health outcomes in this population. Care for adolescent alcohol use is lacking in most pediatric primary care settings (PPC). This project is a pragmatic comparative effectiveness and implementation study that employs a superiority, two-arm, randomized, prospective, observer-blinded, controlled trial design to compare the effectiveness of a patient-centered brief motivational interviewing-based alcohol intervention (BMAI) alone to the same BMAI augmented with adjunctive smartphone app-delivered mindfulness training (MT) for alcohol use in adolescents receiving primary care in PPC clinics across a regional health network. Main effectiveness outcomes will be alcohol use and alcohol related problems assessed over a one-year follow-up period. Implementation outcomes and mediators and moderators of intervention response will also be examined as part of the study.

DETAILED DESCRIPTION:
Alcohol use is prevalent in U.S. adolescents and contributes to adverse health outcomes in this population. Over the past decade, screening, brief intervention, and referral to treatment (SBIRT) has become the primary model for addressing alcohol problems in US adolescents in pediatric healthcare settings. However, uptake and fidelity of SBIRT vary widely in real world settings and barriers to implementing effective brief interventions are common. Standard brief alcohol interventions (BAIs) have predominantly applied motivational interviewing (MI) and feedback techniques to target alcohol and other drug use in adolescents. There is a need to expand BAI options for youth who do not respond to these standard approaches. One intervention approach with growing societal interest and emerging evidence for efficacy in adolescent alcohol and other drug use is mindfulness training (MT). This project will compare two types of evidenced-based care for alcohol use in adolescents recruited from 13 pediatric primary care clinics in a regional health system. The interventions will be a patient-centered brief motivational interviewing-based alcohol intervention (BMAI) delivered by PPC clinicians as part of routine care, and BMAI in combination with smartphone app-delivered mindfulness training (BMAI+ MT).

The project is a pragmatic effectiveness and implementation study that employs a superiority, two-arm, randomized, prospective, observer-blinded, controlled trial design to compare the effectiveness of BMAI alone vs. BMAI augmented with adjunctive smartphone app-delivered MT on alcohol outcomes over a one-year follow-up period. The investigators will use the well-established standard BMAI adapted from the Provider Guide: Adolescent SBIRT Using the Screening to Brief Intervention Car, Relax, Alone, Forget, Friends, Trouble (S2BI-CRAFFT) Screening Tool, an evidence-based brief intervention for alcohol use in youth, and the widely disseminated Healthy Minds Program (HMP) smartphone meditation/mindfulness app which is freely available, science-based, and has shown feasibility and efficacy for reducing stress in youth populations. These interventions which combine elements of face-to-face +/- digital delivery and MI +/- MT will be tested in PPC clinics throughout the Johns Hopkins Medical Institute (JHMI) healthcare network which primarily serves racially/ethnically diverse population of urban and suburban youth in the greater Baltimore/Washington region that has a high proportion of minoritized youth.

The project seeks to answer the following three research questions:

Comparative effectiveness outcomes: What is the relative effectiveness of face-to-face clinician-administered BMAI with vs. without adjunctive app-delivered MT with the HMP app for alcohol using youth in PPC settings? Does supplementing clinician-administered BMAI with app-delivered MT result in superior outcomes in the form of reduced alcohol use and problems for this population or subgroups of the population?

Implementation outcomes: What are the patient and stakeholder perspectives, experiences, and preferences related to delivering BAI with these different components? What are the barriers and facilitators to delivering these BAI in PPC settings and for the diverse patient population served?

Heterogeneity of treatment effect (HTE) outcomes: How do baseline factors such as clinical severity, comorbid psychiatric symptoms and conditions, Socio-economic status (SES), sex, race, ethnicity, caregiver involvement, treatment preference, organization and clinical site readiness, and level of SBIRT integration at PPC clinic sites moderate outcomes across comparator interventions? How do changes in factors that may be mechanism of behavioral change (MOBC) for the different interventions (e.g. 'intrinsic' motivation to quit/reduce drinking, self-efficacy, and goal commitment for MI and mindfulness, anxiety, depression, impulsivity, and self-regulation for MT) and degree of engagement with intervention components (e.g., no. of sessions attended, time spent and no. of MT exercises completed, application of mindfulness in real-life settings) mediate outcomes across comparator interventions? Which patient subgroups benefit the most from which specific mindfulness and motivational BAI components?

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old
* Receiving pediatric primary care (PPC) services through the Johns Hopkins Medical Institute healthcare network
* Screening positive for moderate or high alcohol use risk as indicated by a S2BI score (i.e., showing any monthly alcohol use in the past 12 months)
* Able to speak, understand, and read in English or Spanish
* Able to provide assent, and receiving parental consent/permission to participate.

Exclusion Criteria:

* Severe medical or psychiatric condition (e.g., behavioral dysregulation, psychopathology, or cognitive impairment that in the judgement of study or PPC provider may make participation hazardous [e.g., psychosis, homicidality, active suicidality, mania])
* Intellectual Disability (self-, caregiver-, or PPC-reported, or PPC-documented)
* Current or recent specialty substance use disorder treatment in the past 6 months
* Demonstrated current physiological alcohol withdrawal requiring urgent inpatient referral in the judgement of study or PPC physician
* Reported regular opioid, benzodiazepine, or cocaine use (> weekly) or history of opioid, benzodiazepine, or cocaine overdose in the past 6 months
* Previous experience with a mindfulness-based intervention in the past 12 months
* Current regular meditation practice (> 30 min/day for > 5 days avg. over 30 days prior to screening).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use (total standard drinks) in the past 30 days | Baseline, 1, 3, 6, and 12 months
  Alcohol use (total standard drinks) in the past 30 days, measured via Timeline Follow Back (TLFB) calendar method at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.
Acceptability of intervention (adolescent report) assessed by the Client Satisfaction Questionnaire-Patient Report | Month 2
  Adolescent reported acceptability of BMAI and MT intervention components will be assessed via the Client Satisfaction Questionnaire-Patient Report (CSQ-Patient Report) collected at month 2. CSQ Patient Report scale ranges from 0 to 32 with higher scores indicating greater satisfaction with the intervention.
Acceptability of intervention (caregiver report) assessed by the Client Satisfaction Questionnaire-Caregiver Report | Month 2
  Caregiver reported acceptability of BMAI and MT components will be assessed via the Client Satisfaction Questionnaire-Caregiver Report (CSQ-Caregiver Report) at month 2. CSQ Caregiver Report scale ranges from 0 to 32 with higher scores indicating greater satisfaction with the intervention.
Acceptability of intervention (provider report) assessed by the Provider Satisfaction Questionnaire | month 3, and month 12
  Provider reported acceptability of BMAI and MT components will be assessed via the Provider Satisfaction Questionnaire (PSQ), an adapted form of the Client Satisfaction Questionnaire at month 3 and month 12. PSQ scale ranges from 0 to 32 with higher scores indicating greater satisfaction with the intervention.
Intervention experiences, perspectives, and preferences (adolescent report) assessed by qualitative interview | Month 2
  Adolescent reported personal experiences, perspectives, and preferences related to BMAI and MT components, assessed via qualitative semi-structured interviews obtained from adolescent participants at 2 months. Themes and sub-themes using a grounded theory, inductive approach will be used to identify patient experience with the study arms and interventions.
Intervention experiences, perspectives, and preferences (caregiver report) assessed by qualitative interview | Month 2
  Caregiver reported personal experiences, perspectives, and preferences related to BMAI and MT components, assessed via qualitative semi-structured interviews obtained from caregiver's of adolescent participants at 2 months. Themes and sub-themes using a grounded theory, inductive approach will be used to identify patient experience with the study arms and interventions.
Intervention experiences, perspectives, and preferences (provider report) assessed by qualitative interview | month 3, and month 12
  Provider reported personal experiences, perspectives, and preferences related to BMAI and MT components, assessed via qualitative semi-structured interviews obtained from pediatric primary care (PPC) providers obtained at months 3 and 12. Themes and sub-themes using a grounded theory, inductive approach will be used to identify patient experience with the study arms and interventions.
Implementation barriers and facilitators for SBIRT and BMAI (provider report) | Baseline, month 3, and month 12
  Provider reported barriers and facilitators related to implementation of BMAI intervention and screening brief intervention and referral to treatment (SBIRT) framework, assessed using items about perceived barriers and facilitators from the SBIRT provider questionnaire obtained from PPC clinicians at baseline, month 3, and month 12. The SBIRT provider questionnaire includes questions on substance use screening, brief intervention, and SBIRT practices and perceived barriers and facilitators to screening, providing brief interventions, and implementing SBIRT in their PPC office setting. Number of barriers, number of facilitators, and percentage of providers reporting specific types of barriers and facilitators will be serve as the implementation outcome.
Percentage of providers reporting barriers and facilitators (provider report) | Baseline, month 3, and month 12
  Percentage of providers reporting specific types of barriers and facilitators will serve as the implementation outcome.

SECONDARY OUTCOMES:
Heavy episodic drinking (HED) days in the past 30 days | Baseline, 1, 3, 6, and 12 months
  Heavy episodic drinking days in the past 30 days (defined as number of days in the past 30 days where participant consumed > 5 drinks for male and > 4 drinks for female participants in single session), measured via TLFB calendar method at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.
Cannabis use days in the past 30 days | Baseline, 1, 3, 6, and 12 months
  Cannabis/ tetrahydrocannabinol (THC) product use days in the past 30 days, measured via TLFB calendar method at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.
Tobacco/nicotine use days in the past 30 days | Baseline, 1, 3, 6, and 12 months
  Tobacco/nicotine product use days in the past 30 days, measured via TLFB calendar method at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.
Other drug use days in the past 30 days | Baseline, 1, 3, 6, and 12 months
  Other drug use days in the past 30 days (defined as number of days in the past 30 days where drugs other than alcohol, cannabis, tobacco/nicotine were used), measured via TLFB calendar method at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.
Alcohol-related problem severity assessed by the Alcohol Use Disorders Identification Test | Baseline, 1, 3, 6, and 12 months
  Alcohol-related problem severity measured via the Alcohol Use Disorders Identification Test consumption questions (AUDIT-C) at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The AUDIT-C consists of 3 items assessing typical drinking frequency, typical drinking quantity, and frequency of heavy episodic drinking, each scored from 0 to 4. The AUDIT-C composite score has a scale that ranges from 0 to 12 with higher scores indicating greater alcohol problem severity. A total AUDIT-C score > or equal to 3 has a good sensitivity and specificity for detecting alcohol use problems in adolescents.
Recent Alcohol Consumption (past 7 days) | Baseline, 1, 3, 6, and 12 months
  Recent alcohol consumption (defined as total number of standard drinks in the past 7 days), measured via TLFB calendar method at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.
Alcohol-related consequences assessed by the Short Index of Problems | Baseline, 1, 3, 6, and 12 months
  Alcohol-related consequences assessed with the Short Index of Problems (SIP) related to alcohol consumption at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The SIP consists of 17 questions each scored from 0 to 3. The scale ranges from 0 to 51 with higher scores indicating greater occurrence of alcohol related negative consequences.
Emergency health service utilization | Baseline, 1, 3, 6, and 12 months
  Emergency health service utilization (defined as the number of visits to the emergency room for health treatment), measured via 1-item on emergency department visits from The Economic Form-90 at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.
Quality of Life (QOL) as assessed by the Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline, 1, 3, 6, and 12 months
  Quality of Life (QOL) assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) pediatric global health (PGH-7) index at five time points (baseline and 1, 2, 3, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups.The PROMIS PGH-7 index consists of 7 questions each scored from 1 to 5. The scale ranges from 7 to 35 with higher scores indicating greater QOL and general health.

OTHER OUTCOMES:
Drinking to Cope (DTC) with negative emotions assessed by the 5 item Coping Subscale | Baseline, 1, 3, 6, and 12 months
  Drinking to Cope (DTC) with negative emotions assessed with the 5-item Coping Subscale of the Drinking Motives Questionnaire-Revised (DMQ-R) at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The DTC subscale ranges from 5 to 25 with higher scores indicating greater coping motives for alcohol use.
Alcohol Cravings assessed by the 5 item Penn Alcohol Craving scale | Baseline, 1, 3, 6, and 12 months
  Alcohol cravings assessed with the 5-Item Penn Alcohol Craving Scale (PACS) at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The PACS scale ranges from 0 to 30 with higher scores indicating greater cravings for alcohol use in the past week.
Dispositional Mindfulness assessed by the10 item Child and Adolescent Mindfulness Measure | Baseline, 1, 3, 6, and 12 months
  Dispositional Mindfulness assessed with the 10-Item Child and Adolescent Mindfulness Measure (CAAM), at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The CAAM scale ranges from 0 to 40 with higher scores indicating greater levels of dispositional mindfulness. Dispositional mindfulness at baseline and change in dispositional mindfulness during/following treatment will be examined as potential moderators and mediators of BMAI vs. BMAI + MT intervention effects on alcohol outcomes, respectively.
Mindfulness Practice assessed by Applied Mindfulness Process Scale | Baseline, 1, 3, 6, and 12 months
  Mindfulness practice (defined as use of mindfulness skills in day-to-day life) assessed with the Applied Mindfulness Process Scale (AMPS), at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The AMPS scale ranges from 0 to 60 with higher scores indicating greater application of mindfulness skills in daily life coinciding with mindfulness practice. Mindfulness practice will be examined as a potential mediator of BMAI vs. BMAI + MT intervention effects on alcohol outcomes.
Healthy Mind Program (HMP) App Usage | 1, 3, 6, and 12 months
  Healthy Minds Program (HMP) mindfulness app usage data on the number of completed HMP practices/exercises, modules used, will be collected from each participant in the BMAI + MT group. This app usage data will be examined as a potential mediator of BMAI vs. BMAI + MT intervention effects on alcohol outcomes.
Healthy Mind Program (HMP) App Usage (time spent) | 1, 3, 6, and 12 months
  Healthy Minds Program (HMP) mindfulness app usage data on the time spent (minutes) using the HMP app will be collected from each participant in the BMAI + MT group. This app usage data will be examined as a potential mediator of BMAI vs. BMAI + MT intervention effects on alcohol outcomes.
Healthy Mind Program (HMP) App Usage (days of usage) | 1, 3, 6, and 12 months
  Healthy Minds Program (HMP) mindfulness app usage data on the days spent using the HMP app will be collected from each participant in the BMAI + MT group. This app usage data will be examined as a potential mediator of BMAI vs. BMAI + MT intervention effects on alcohol outcomes.
Healthy Mind Program (HMP) Proportion of participant usage | 1, 3, 6, and 12 months
  Aggregate app use data (proportion of participants in the BMAI + MT group completing 50%, 75%, and 100% of HMP exercises and modules) will serve as an index of app uptake and engagement for the study.
Depression assessed by the Patient Health Questionnaire for Adolescents | Baseline, 1, 3, 6, and 12 months
  Depression assessed with the Patient Health Questionnaire for Adolescents (PHQ-9-A) at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The PHQ-9-A scale ranges from 0 to 27 with higher scores indicating higher depression severity. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe depression, respectively. A total PHQ-9-A score > 10 has a good sensitivity and specificity for Major Depressive Disorder in adolescents in PPC. Depression at baseline and change in depression severity during/following treatment will be examined as potential moderators and mediators of BMAI vs. BMAI + MT intervention effects on alcohol outcomes.
Anxiety assessed by the Generalized Anxiety Disorder Scale | Baseline, 1, 3, 6, and 12 months
  Anxiety assess with the Generalized anxiety disorder (GAD-7) scale at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The GAD-7 scale ranges from 0 to 21 with higher scores indicating higher anxiety severity. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. A total GAD-7 score > 10 has a good sensitivity and specificity for Generalized Anxiety Disorder among adolescents in PPC. Anxiety at baseline and change in anxiety severity during/following treatment will be examined as potential moderators and mediators of BMAI vs. BMAI + MT intervention effects on alcohol outcomes, respectively.
Impulsivity assessed by the Short-version of the Urgency Pre-meditation Perseverance Sensation Seeking Positive Urgency | Baseline, 1, 3, 6, and 12 months
  Impulsivity assessed with the Short-Version of the Urgency-Premeditation-Perseverance-Sensation Seeking-Positive Urgency (UPPS-P) negative urgency subscale at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The negative urgency subscale of the UPPS-P consists of 4 items scored from 1 to 4. The subscale ranges from 4 to 16 with higher scores indicating a greater tendency to act impulsively or rashly when experiencing negative emotions. Impulsivity at baseline and change in impulsivity during/following treatment will be examined as potential moderators and mediators of BMAI vs. BMAI + MT intervention effects on alcohol outcomes, respectively.
Emotion Regulation assessed by the16 item Brief Version of the Difficulties in Emotion Regulation Scale | Baseline, 1, 3, 6, and 12 months
  Emotion regulation assessed with the 16-item Brief Version of the Difficulties in Emotion Regulation Scale (DERS-16) at five time points (baseline and 1, 3, 6, and 12 months) over a one year follow-up period, compared between BMAI and BMAI + MT groups. The DERS-16 scale ranges from 16 to 80 with higher scores indicating greater levels of emotion dysregulation. Emotion regulation at baseline and change in emotion regulation during/following treatment will be examined as potential moderators and mediators of BMAI vs. BMAI + MT intervention effects on alcohol outcomes, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Hammond, MD, PhD, Principal Investigator — Johns Hopkins University; Hoover Adger, MD, MPH, MBA, Study Director — Johns Hopkins University
Locations (13):
- United States (13):
  - Johns Hopkins Community Physicians, Remington, Baltimore, Maryland
  - Johns Hopkins Bayview Pediatrics (Baltimore Medical System, Yard 56), Baltimore, Maryland
  - Johns Hopkins Community Physicians, Canton Crossing, Baltimore, Maryland
  - Harriet Lane Clinic, Baltimore, Maryland
  - Johns Hopkins University Center for Adolescent and Young Adult Health, Baltimore, Maryland
  - Johns Hopkins Community Physicians, Water's Edge, Belcamp, Maryland
  - Johns Hopkins Community Physicians, Bowie, Bowie, Maryland
  - Johns Hopkins Community Physicians, Howard County Pediatrics, Columbia, Maryland
  - Johns Hopkins Community Physicians, Glen Burnie, Glen Burnie, Maryland
  - Johns Hopkins Community Physicians, Hagerstown, Hagerstown, Maryland
  - Johns Hopkins Community Physicians, White Marsh Pediatrics, Nottingham, Maryland
  - Johns Hopkins Community Physicians, Odenton Medical, Odenton, Maryland
  - Johns Hopkins Community Physicians, Rockville Pediatrics, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No